CLINICAL TRIAL: NCT04949711
Title: Impacts of Subsidized Ridesharing on Drunk Driving, Alcohol Consumption, and Mobility
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, Christopher Morrison, Assistant Professor of Epidemiology, Columbia University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: AAAT0912; 1R01AA029112-01 (NIH)
Record Dates: First submitted 2021-06-25; First posted 2021-07-02 (Actual); Last update posted 2025-04-13 (Actual); Status verified 2025-04

CONDITIONS: Driving Drunk; Alcohol Drinking
Keywords: Drunk driving; Ridesharing; Alcohol Drinking; Driving under the influence (DUI)
MeSH Terms: conditions — Driving Under the Influence; Alcohol Drinking

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Experimental): Participants will be asked to complete 3 surveys over 2 weeks to collect in information on their alcohol use and about themselves, and receive ridesharing vouchers.
  Interventions: Behavioral: ridesharing voucher
- Control (Sham Comparator): Participants will be asked to complete 3 surveys over 2 weeks to collect in information on their alcohol use and about themselves, and receive online shopping voucher.
  Interventions: Behavioral: online shopping voucher

INTERVENTIONS:
Behavioral: ridesharing voucher — Ridesharing vouchers will be given for completing each of the online surveys, for a possible total of $80 if you complete all three surveys. You will be paid with electronic vouchers that will be sent to your cell phone.
  Other Names: Uber voucher
  Arms: Intervention
Behavioral: online shopping voucher — Online shopping vouchers will be given for completing each of the online surveys, for a possible total of $80 if you complete all three surveys. You will be paid with electronic vouchers that will be sent to your cell phone.
  Other Names: Amazon voucher
  Arms: Control

SUMMARY:
The purpose of this research study is to understand people's alcohol use in public places and their risks for harm. The overall goal of this study is to test the effects of subsidized ridesharing as an intervention to reduce self-reported alcohol-impaired driving, along with alcohol consumption and changes to mobility.

DETAILED DESCRIPTION:
Motor vehicle crashes are the leading cause of death for people aged 13-25 years in the US, and approximately 31% of all fatal crashes involved some alcohol use. Several peer-reviewed studies have found that ridesharing was associated with fewer alcohol-involved crashes and DUI arrests. Theories of behavioral economics provide a clear theoretical mechanism by which ridesharing will reduce alcohol-involved motor vehicle crashes compared to other private transportation. However, while ridesharing may be an effective intervention to reduce alcohol-involved crashes, it may simultaneously increase alcohol consumption. This study will assess the impacts of subsidized ridesharing on impaired driving, alcohol consumption, and mobility. Participants will be randomized to either receive a rideshare voucher or an online shopping voucher, and effects on alcohol impaired driving and alcohol consumption will be measured. A GPS sub-group will use a custom smartphone application for GPS tracking to measure mobility.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 21 years old
* Reside in a study city
* Have a driver's license
* Have access to a motor vehicle
* Have consumed alcohol in a bar in the last 30 days
* Own a smartphone
* Read English

Exclusion Criteria:

* Non-English speaking participants

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 7034 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2025-03-14 (Actual); Study Completion 2025-04-04 (Actual)

PRIMARY OUTCOMES:
Change in the alcohol impaired driving incidents | Baseline, 1 week follow-up, 2 week follow-up
  Participants will provide two self-reported measures of impaired driving by indicating whether they "drove after drinking any alcohol" (driving after drinking) and "drove after drinking too much alcohol to drive safely" (driving while intoxicated) for each day during the previous 7 days.

SECONDARY OUTCOMES:
Change in number of days in alcohol consumption | Baseline, 1 week follow-up, 2 week follow-up
  Participants will be asked to state the number of drinks consumed on each day for the 7 previous days, and their responses will be used to calculate the frequency (defined as the number of drinking days) and the continued volume (defined as total number of drinks consumed after 1 drink on a drinking day) of drinking.
Average frequency of trips to alcohol outlets | Day 3 to Day 17 of study
  Participants enrolled in the GPS sub-sample will be tracked and GPS records will be used measure exposure to alcohol outlets and mobility.
Average duration of trips to alcohol outlets | Day 3 to Day 17 of study
  Participants enrolled in the GPS sub-sample will be tracked and GPS records will be used measure exposure to alcohol outlets and mobility.
Change in The Drinker Inventory of Consequences Score | Baseline, 1 week follow-up, 2 week follow-up
  The Drinker Inventory of Consequences is a 45-item measure of alcohol-related consequences on which higher scores reflect greater alcohol consequences. It measures harms related to alcohol consumption within 5 sub-scales: physical consequences, intrapersonal consequences, social responsibility consequences, interpersonal consequences, and impulse control consequences.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Morrison, PhD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Irving Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Data from the study will be submitted and shared with NIAAA Data Archive (NIAAADA), a data repository housed within the NIMH Data Archive (NDA).
Supporting Information: Analytic Code
Time Frame: Data will become available March 2028, 2 years after the end of the project, as designated by NIAAADA policy.
Access Criteria: Study data can be accessed on the NIAAADA website: https://nda.nih.gov/niaaa/getting-data For access to individual-level data, researchers will need to receive authorization from NIAAA by completing the NDA Data Access Request (DAR).
URL: https://nda.nih.gov/niaaa